CLINICAL TRIAL: NCT05430503
Title: Lung Diffusing Capacities for Nitric Oxide and Carbon Monoxide in Long COVID With Dyspnea at Rest and After Mild Exercise
Brief Title: Long COVID and Post-exertional Pulmonary Diffusion
Acronym: Long_COVID_Ex
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Giovanni Barisione, Chief, Respiratory Pathophysiology, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Other Study IDs: Long_COVID_Exer_DLNO_DLCO
Record Dates: First submitted 2022-06-19; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Long COVID; Breathlessness; Exercise Intolerance; Alveolar Lung Disease; Pulmonary Gas Exchange
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Dyspnea | interventions — Lung Volume Measurements; Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long COVID: Caucasian subjects with a history of SARS CoV-2 infection confirmed by nasopharyngeal swab with real-time polymerase-chain reaction were included in the study. They were referred to investigators' pulmonary function laboratory after being tested negative for SARS-CoV-2, because of dyspnea, fatigue, and exercise intolerance persisting or occurring at least 3 months after the COVID-19 acute phase and lasting ≥2 months.
  Interventions: Diagnostic Test: Lung volumes, spirometry and standard single-breath DLCO were measured at rest while combined DLNO and DLCO were measured at rest and post-exercise
- Healthy controls: Anthropometrically-matched healthy subjects, without history of COVID-19 and vaccinated against SARS-CoV-2 infection.
  Interventions: Diagnostic Test: Lung volumes, spirometry and standard single-breath DLCO were measured at rest while combined DLNO and DLCO were measured at rest and post-exercise

INTERVENTIONS:
Diagnostic Test: Lung volumes, spirometry and standard single-breath DLCO were measured at rest while combined DLNO and DLCO were measured at rest and post-exercise — DLNO and DLCO were measured at rest and 5-10 s after a bout of treadmill exercise simulating usual walking

SUMMARY:
Aim of investigators was to study whether abnormalities of lung diffusing capacity for nitric oxide (DLNO) and carbon monoxide (DLCO) in long COVID may have a clinical impact in relation to exercise intolerance.

DETAILED DESCRIPTION:
Prolonged recovery from acute coronavirus disease 2019 (long COVID) is characterized in about 30% of subjects from breathlessness and fatigue also during daily activities often associated to decreased lung diffusing capacity for carbon monoxide (DLCO) at rest. Aim of investigators was to study whether abnormalities of lung diffusing capacity for nitric oxide (DLNO) and DLCO in long COVID may have a clinical impact in relation to exercise intolerance. Combined DLNO and DLCO were simultaneously measured at rest and immediately after a short bout of treadmill walking in 32 dyspneic subjects ≥3 months after the COVID-19 acute phase. A group of healthy subjects served as a control group.

ELIGIBILITY:
Inclusion Criteria:

* History of dyspnea, fatigue, and exercise intolerance persisting or occurring at least 3 months after the COVID-19 acute phase and lasting ≥2 months.

Exclusion Criteria:

* History of diseases potentially causing dyspnea or affecting pulmonary gas transport, i.e., bronchial asthma, lung bullous disease, chronic obstructive pulmonary disease, pulmonary interstitial fibrosis or vasculitis, hematological diseases, systemic collagen diseases, congestive heart failure, liver or renal diseases, and morbid obesity.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Caucasian subjects with a history of SARS CoV-2 infection confirmed by nasopharyngeal swab with real-time polymerase-chain reaction. They were referred to our pulmonary function laboratory after being tested negative for SARS-CoV-2, because of dyspnea, fatigue, and exercise intolerance persisting or occurring at least 3 months after the COVID-19 acute phase and lasting ≥2 months.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Combined DLNO and DLCO changes after mild exercise | through study completion, an average of 6 months
  pulmonary gas exchange abnormalities in dyspneic long COVID subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Policlinico San Martino IRCCS - S.S. Fisiopatologia Respiratoria, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided